CLINICAL TRIAL: NCT03751696
Title: Coaching Intervention to Improve Mental Well-being of Community Women Who Are At-risk of Common Mental Disorders in Hong Kong: A Pilot Randomized Controlled Trials
Brief Title: Coaching Intervention in Women At-risk of Common Mental Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Eric Y.H. Chen, Chair Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CoachingRCT
Record Dates: First submitted 2018-11-10; First posted 2018-11-23 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Common Mental Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group coaching (Experimental): There will be a total of 4 sessions of group coaching intervention within 8 weeks. Each session is in a group of 5-6 women and lasts for approximately 1-1.5 hours. The sessions will be conducted by experienced social workers online.
  Interventions: Behavioral: Group Coaching
- SMS Self-help tips (Active Comparator): The participants in the control group will receive four self-help tips on mental well-being on the same schedule as the group coaching group.
  Interventions: Behavioral: SMS self-help tips

INTERVENTIONS:
Behavioral: Group Coaching — 4 sessions of 1-1.5-hour group coaching intervention within 8 weeks
  Arms: Group coaching
Behavioral: SMS self-help tips — 4 mental well-being tips through sms within 8 weeks
  Arms: SMS Self-help tips

SUMMARY:
This study aims to provide preventative intervention to 60 women who are at risk of common mental disorders in Hong Kong.

DETAILED DESCRIPTION:
Participants will be recruited through the following routes: 1) by our partner non-governmental organizations, 2) by our research team through community outreach or training activities, 3) online screening tool, and 4) referral from organizations that provide service to women (e.g., Maternal and Child Health Clinics of Department of Health). Eligible subjects with informed consent provided will be randomly assigned to coaching group or SMS self-help tips. To test the effectiveness of the provided intervention programs, symptoms assessments and data collection on demographics and psychosocial data will be carried out during baseline, immediately, and 3 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Able to understand Cantonese and read/write Chinese
* With subsyndromal or minor depressive symptoms indicated by
* Depression subscale of Depression, Anxiety and Stress Scale (DASS) score 10-20 or
* Edinburgh Postnatal Depression Scale (EPDS) scores 10-13

Exclusion Criteria:

* A positive response in items about suicidal thoughts if applicable ("Yes, quite often" and "sometimes" in EPDS) (These participants will be referred to suicidal management)
* Those mental conditions that require other treatment priorities (e.g., suicidal risk, substance abuse, current or past episodes of psychotic disorder, personality disorders)
* Those medical conditions that severely limit participation, comprehension, or adherence to treatment (e.g., epilepsy, dementia, terminal medical illness)
* Those who are receiving structured psychotherapy or counseling

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult women
Enrollment: 60 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | immediate post-intervention
  Measured by the depression subscale of the Depression, Anxiety and Stress Scale
Anxiety symptoms | immediate post-intervention
  Measured by the anxiety subscale of the Depression, Anxiety and Stress Scale

SECONDARY OUTCOMES:
Depressive symptoms | 3-month post intervention
  Measured by the depression subscale of the Depression, Anxiety and Stress Scale (DASS). The subscale consists of 7 questions, each responses range from 0 (not applicable) to 3 (the most applicable). The higher score represents more severe depressive symptoms.
Anxiety symptoms | 3-month post intervention
  Measured by the anxiety subscale of the Depression, Anxiety and Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Eric YH Chen, MD, Study Director — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No